CLINICAL TRIAL: NCT07061314
Title: Comparison of Lower Limb COP and Muscle Activation During Single-Leg Deadlift Using Elastic and Inelastic Barbells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Busan University of Foreign Studies (Other)
Responsible Party: Principal Investigator, Ji Hwan Jeong, Principal Investigator, Busan University of Foreign Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUFS-SLDL-2025
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Control; Functional Training; Lower Limb Stability
Keywords: Single-Leg Deadlift; elastic barbell; inelastic barbell; sports rehabilitation; neuromuscular control

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Group Crossover (Experimental): Participants will perform single-leg deadlifts under two loading conditions: an elastic barbell and an inelastic barbell. Each condition will be tested at three different movement speeds (normal, fast, and power) in randomized order. Each participant completes all conditions as part of a within-subject repeated measures design
  Interventions: Device: Elastic Barbell; Device: Inelastic Barbell

INTERVENTIONS:
Device: Elastic Barbell — A flexible plastic barbell that creates top-down perturbations during movement. Participants perform single-leg deadlifts using this elastic bar at three different speeds: normal (2 sec), fast (1 sec), and power (as fast as possible). The bar is loaded to 30% of the participant's estimated 1RM.
Device: Inelastic Barbell — A standard rigid steel barbell with no elasticity. Participants perform single-leg deadlifts using this barbell under the same speed conditions and loading parameters as the elastic barbell.

SUMMARY:
This study aims to investigate the effects of barbell type (elastic vs. inelastic) and lifting speed on lower limb balance and muscle activation during the Single-Leg Deadlift (SLDL) exercise. Using a randomized crossover design, healthy adults performed SLDL at three different movement speeds while center of pressure (COP) and electromyographic (EMG) responses were measured. The study seeks to determine whether elastic barbells, which create top-down perturbations, enhance neuromuscular control and postural stability more effectively than traditional inelastic barbells.

DETAILED DESCRIPTION:
This randomized clinical trial examines how barbell type and movement speed affect lower limb stability and muscle activation during Single-Leg Deadlift (SLDL) exercises. The intervention compares elastic barbells-designed to generate upper-limb-initiated dynamic perturbations-to conventional inelastic barbells. Twenty-seven healthy adults with prior resistance training experience participated in the study. All participants performed SLDL using both barbell types across three speeds: normal (2 seconds), fast (1 second), and power (as fast as possible).

Center of Pressure (COP) data were recorded using a force platform to assess anterior-posterior (AP) and medial-lateral (ML) sway. Surface electromyography (EMG) was collected from eight lower limb muscles to evaluate neuromuscular responses. Data were analyzed using two-way repeated measures ANOVA.

The findings revealed that elastic barbells significantly reduced COP displacement and increased activation in the gluteus medius, biceps femoris, semitendinosus, and gastrocnemius muscles-particularly at high movement speeds. These results suggest that elastic barbells may improve dynamic stability and neuromuscular coordination, offering potential applications in sports rehabilitation and unilateral training programs.

ELIGIBILITY:
Inclusion Criteria:

* No history of musculoskeletal disorders in the past 6 months

At least 1 year of experience in resistance or functional training

Able to perform single-leg deadlift exercise safely

Provided written informed consent

Exclusion Criteria:

* History of lower extremity surgery or major musculoskeletal injury within the past year

Current pain or symptoms in the hip, knee, or ankle joints

Neurological, cardiovascular, or balance disorders

Participation in other conflicting research studies within the last 3 months

Inability to maintain single-leg stance for at least 5 seconds

Presence of skin irritation or condition at electrode placement sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Center of Pressure Displacement - Anterior-Posterior (AP) | During single-leg deadlift task (within single session)
  The range of anterior-posterior (AP) sway displacement (in centimeters) will be measured using a force platform (AMTI OR6). Participants perform SLDL under both barbell conditions at three different movement speeds. Lower values indicate greater postural stability.
Center of Pressure Displacement - Medial-Lateral (ML) | During single-leg deadlift task (within single session)
  The range of medial-lateral (ML) sway displacement (in centimeters) will be measured using a force platform (AMTI OR6). The COP variability is analyzed as an indicator of dynamic balance control.
Muscle Activation of Lower Limb Muscles (%MVIC) | During single-leg deadlift task (within single session)
  Surface electromyography (EMG) will be used to measure muscle activation in eight lower limb muscles during single-leg deadlifts under elastic and inelastic barbell conditions at three movement speeds (normal, fast, power). The muscles assessed include gluteus medius, rectus femoris, vastus medialis, vastus lateralis, biceps femoris, semitendinosus, gastrocnemius, and tibialis anterior.
  EMG signals will be processed using RMS and normalized to maximum voluntary isometric contraction (%MVIC). Increased %MVIC indicates higher neuromuscular demand under perturbation.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hwan Jeong, MSc, Principal Investigator — Department of Sports and Health Convergence
Locations (1):
- Busan University of Foreign Studies, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared via Figshare. The data will include demographic information, raw data from the assessments, and any other relevant data collected during the study.
Supporting Information: SAP
Time Frame: The data will be available immediately after the publication of the study results and will be accessible for at least 5 years
Access Criteria: The data will be openly available via Figshare without the need for a data access request

REFERENCES:
- [Background] Ditroilo M, O'Sullivan R, Harnan B, Crossey A, Gillmor B, Dardis W, Grainger A. Water-filled training tubes increase core muscle activation and somatosensory control of balance during squat. J Sports Sci. 2018 Sep;36(17):2002-2008. doi: 10.1080/02640414.2018.1431868. Epub 2018 Jan 24. PMID 29364062
- [Background] Saeterbakken AH, Fimland MS. Muscle force output and electromyographic activity in squats with various unstable surfaces. J Strength Cond Res. 2013 Jan;27(1):130-6. doi: 10.1519/JSC.0b013e3182541d43. PMID 22450254
- [Background] Badier M, Guillot C, Lagier-Tessonnier F, Burnet H, Jammes Y. EMG power spectrum of respiratory and skeletal muscles during static contraction in healthy man. Muscle Nerve. 1993 Jun;16(6):601-9. doi: 10.1002/mus.880160605. PMID 8502257
- [Background] Rutherford DJ, Hubley-Kozey CL, Stanish WD. Maximal voluntary isometric contraction exercises: a methodological investigation in moderate knee osteoarthritis. J Electromyogr Kinesiol. 2011 Feb;21(1):154-60. doi: 10.1016/j.jelekin.2010.09.004. PMID 20926310
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Lafond D, Corriveau H, Hebert R, Prince F. Intrasession reliability of center of pressure measures of postural steadiness in healthy elderly people. Arch Phys Med Rehabil. 2004 Jun;85(6):896-901. doi: 10.1016/j.apmr.2003.08.089. PMID 15179642
- [Background] Lopez-de-Celis C, Sanchez-Alfonso N, Rodriguez-Sanz J, Romani-Sanchez S, Labata-Lezaun N, Canet-Vintro M, Aiguade R, Perez-Bellmunt A. Quadriceps and gluteus medius activity during stable and unstable loading exercises in athletes. A cross-sectional study. J Orthop Res. 2024 Feb;42(2):317-325. doi: 10.1002/jor.25680. Epub 2023 Aug 27. PMID 37593805
- [Background] Morrissey MC, Harman EA, Johnson MJ. Resistance training modes: specificity and effectiveness. Med Sci Sports Exerc. 1995 May;27(5):648-60. PMID 7674868
- [Background] Hutchison RE, Caterisano A. Comparison of Peak Ground Reaction Force, Joint Kinetics and Kinematics, and Muscle Activity Between a Flexible and Steel Barbell During the Back Squat Exercise. J Hum Kinet. 2019 Aug 21;68:99-108. doi: 10.2478/hukin-2019-0059. eCollection 2019 Aug. PMID 31531136
- [Background] Glass SC, Wisneski KA. Effect of Instability Training on Compensatory Muscle Activation during Perturbation Challenge in Young Adults. J Funct Morphol Kinesiol. 2023 Sep 15;8(3):136. doi: 10.3390/jfmk8030136. PMID 37754969
- [Background] Mansfield A, Wong JS, Bryce J, Knorr S, Patterson KK. Does perturbation-based balance training prevent falls? Systematic review and meta-analysis of preliminary randomized controlled trials. Phys Ther. 2015 May;95(5):700-9. doi: 10.2522/ptj.20140090. Epub 2014 Dec 18. PMID 25524873
- [Background] Pai YC, Bhatt T, Yang F, Wang E. Perturbation training can reduce community-dwelling older adults' annual fall risk: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1586-94. doi: 10.1093/gerona/glu087. Epub 2014 Jun 24. PMID 24966227
- [Background] Smania N, Corato E, Tinazzi M, Stanzani C, Fiaschi A, Girardi P, Gandolfi M. Effect of balance training on postural instability in patients with idiopathic Parkinson's disease. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):826-34. doi: 10.1177/1545968310376057. PMID 21045119
- [Background] Nairn BC, Sutherland CA, Drake JD. Motion and Muscle Activity Are Affected by Instability Location During a Squat Exercise. J Strength Cond Res. 2017 Mar;31(3):677-685. doi: 10.1519/JSC.0000000000001745. PMID 27930445
- [Background] Drinkwater EJ, Pritchett EJ, Behm DG. Effect of instability and resistance on unintentional squat-lifting kinetics. Int J Sports Physiol Perform. 2007 Dec;2(4):400-13. doi: 10.1123/ijspp.2.4.400. PMID 19171958
- [Background] Behm DG, Anderson KG. The role of instability with resistance training. J Strength Cond Res. 2006 Aug;20(3):716-22. doi: 10.1519/R-18475.1. PMID 16937988
- [Background] Dominguez-Navarro F, Casana J, Perez-Dominguez B, Ricart-Luna B, Cotoli-Suarez P, Calatayud J. Dynamic balance and explosive strength appears to better explain single leg hop test results among young elite female basketball athletes. Sci Rep. 2023 Apr 4;13(1):5476. doi: 10.1038/s41598-023-31178-7. PMID 37016001
- [Background] Gonzalo-Skok O, Tous-Fajardo J, Suarez-Arrones L, Arjol-Serrano JL, Casajus JA, Mendez-Villanueva A. Single-Leg Power Output and Between-Limbs Imbalances in Team-Sport Players: Unilateral Versus Bilateral Combined Resistance Training. Int J Sports Physiol Perform. 2017 Jan;12(1):106-114. doi: 10.1123/ijspp.2015-0743. Epub 2016 Aug 24. PMID 27140680
- [Background] Speirs DE, Bennett MA, Finn CV, Turner AP. Unilateral vs. Bilateral Squat Training for Strength, Sprints, and Agility in Academy Rugby Players. J Strength Cond Res. 2016 Feb;30(2):386-92. doi: 10.1519/JSC.0000000000001096. PMID 26200193
- [Background] Makaruk H, Winchester JB, Sadowski J, Czaplicki A, Sacewicz T. Effects of unilateral and bilateral plyometric training on power and jumping ability in women. J Strength Cond Res. 2011 Dec;25(12):3311-8. doi: 10.1519/JSC.0b013e318215fa33. PMID 22076090
- [Background] Gholami F, Letafatkar A, Moghadas Tabrizi Y, Gokeler A, Rossettini G, Ghanati HA, Schollhorn WI. Comparing the Effects of Differential and Visuo-Motor Training on Functional Performance, Biomechanical, and Psychological Factors in Athletes after ACL Reconstruction: A Randomized Controlled Trial. J Clin Med. 2023 Apr 13;12(8):2845. doi: 10.3390/jcm12082845. PMID 37109182
- [Background] Correa RV, Verhagen E, Resende RA, Ocarino JM. Performance in field-tests and dynamic knee valgus in soccer players psychologically ready and not ready to return to sports after ACL reconstruction. Knee. 2023 Jun;42:297-303. doi: 10.1016/j.knee.2023.04.011. Epub 2023 Apr 27. PMID 37119602
- [Background] van Dyk N, Behan FP, Whiteley R. Including the Nordic hamstring exercise in injury prevention programmes halves the rate of hamstring injuries: a systematic review and meta-analysis of 8459 athletes. Br J Sports Med. 2019 Nov;53(21):1362-1370. doi: 10.1136/bjsports-2018-100045. Epub 2019 Feb 26. PMID 30808663
- [Background] Maniar N, Cole MH, Bryant AL, Opar DA. Muscle Force Contributions to Anterior Cruciate Ligament Loading. Sports Med. 2022 Aug;52(8):1737-1750. doi: 10.1007/s40279-022-01674-3. Epub 2022 Apr 18. PMID 35437711
- [Background] Biscarini A, Benvenuti P, Botti FM, Brunetti A, Brunetti O, Pettorossi VE. Voluntary enhanced cocontraction of hamstring muscles during open kinetic chain leg extension exercise: its potential unloading effect on the anterior cruciate ligament. Am J Sports Med. 2014 Sep;42(9):2103-12. doi: 10.1177/0363546514536137. Epub 2014 Jun 10. PMID 24918112
- [Background] Begalle RL, Distefano LJ, Blackburn T, Padua DA. Quadriceps and hamstrings coactivation during common therapeutic exercises. J Athl Train. 2012 Jul-Aug;47(4):396-405. doi: 10.4085/1062-6050-47.4.01. PMID 22889655
- [Background] Llurda-Almuzara L, Perez-Bellmunt A, Lopez-de-Celis C, Aiguade R, Seijas R, Casasayas-Cos O, Labata-Lezaun N, Alvarez P. Normative data and correlation between dynamic knee valgus and neuromuscular response among healthy active males: a cross-sectional study. Sci Rep. 2020 Dec 2;10(1):17206. doi: 10.1038/s41598-020-74177-8. PMID 33268811
- [Background] Llurda-Almuzara L, Perez-Bellmunt A, Labata-Lezaun N, Lopez-de-Celis C, Canet-Vintro M, Cadellans-Arroniz A, Moure-Romero L, Aiguade-Aiguade R. Relationship between lower limb EMG activity and knee frontal plane projection angle during a single-legged drop jump. Phys Ther Sport. 2021 Nov;52:13-20. doi: 10.1016/j.ptsp.2021.07.007. Epub 2021 Jul 29. PMID 34365085
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026
- [Background] Distefano LJ, Blackburn JT, Marshall SW, Padua DA. Gluteal muscle activation during common therapeutic exercises. J Orthop Sports Phys Ther. 2009 Jul;39(7):532-40. doi: 10.2519/jospt.2009.2796. PMID 19574661
- [Background] Mo RCY, Ngai DCW, Ng CCM, Sin KHS, Luk JTC, Ho IMK. Effects of loading positions on the activation of trunk and hip muscles during flywheel and dumbbell single-leg Romanian deadlift exercises. Front Physiol. 2023 Nov 29;14:1264604. doi: 10.3389/fphys.2023.1264604. eCollection 2023. PMID 38093908
- [Background] Diamant W, Geisler S, Havers T, Knicker A. Comparison of EMG Activity between Single-Leg Deadlift and Conventional Bilateral Deadlift in Trained Amateur Athletes - An Empirical Analysis. Int J Exerc Sci. 2021 Apr 1;14(1):187-201. doi: 10.70252/MVFY4610. eCollection 2021. PMID 34055137